CLINICAL TRIAL: NCT03006276
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy, Tolerability, and Safety Study of DFN-15 in Episodic Migraine With or Without Aura
Brief Title: Efficacy, Tolerability, and Safety Study of DFN-15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFN-15-CD-007
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFN-15 Active (Experimental): DFN-15 Active
  Interventions: Drug: DFN-15 Active
- DFN-15 Placebo (Placebo Comparator): DFN-15 Placebo
  Interventions: Other: DFN-15 Placebo

INTERVENTIONS:
Drug: DFN-15 Active
  Other Names: Celecoxib Oral Solution
  Arms: DFN-15 Active
Other: DFN-15 Placebo
  Arms: DFN-15 Placebo

SUMMARY:
Efficacy, Tolerability, and Safety of DFN-15 in episodic migraine with or without aura, being conducted at multiple centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. A history of episodic migraine, who experience 2 to 8 migraine attacks per month for at least the past 12 months, with no more than 14 headache days per month, and with 48 hours of headache-free time between migraine attacks.
2. Patients who have migraine with or without aura with onset before age 50 years
3. Report usual migraine pain of 2 (moderate) or 3 (severe) on headache pain severity scale without treatment.
4. Subjects who are willing and able to:

   1. Evaluate and record pain, migraine symptoms, and study drug effectiveness information in real-time using a subject eDiary for the duration of the study;
   2. Record each instance of the use of study drug and rescue medication in real-time using a subject eDiary for the duration of the study;
   3. Comply with all other study procedures and scheduling requirements.

Exclusion Criteria:

1. Minors, even if they are in the specified study age range
2. Medication overuse:

   1. Opioids greater than or equal to 10 days during the 90 days prior to screening
   2. Combination medications (e.g., Fiorinal®) greater than or equal to 10 days during the 90 days prior to screening (applies only if includes opioid and/or barbiturate)
   3. Nonsteroidal Anti-inflammatory Drugs or other simple medications greater than 14 days a month during the 90 days prior to screening
   4. Triptans or ergots greater than or equal to 10 days a month during the 90 days prior to screening
3. Treated with onabotulinumtoxin A (Botox®) for migraine within 4 months prior to screening. (If treated for cosmetic reasons, subjects may be included).
4. Current treatment with antipsychotics or use of antipsychotics within 30 days prior to randomization.
5. Patients who have received treatment with an investigational drug or device within 30 days of randomization, or participated in a central nervous system clinical trial within 2 months prior to randomization
6. Patients with positive screening test for human immunodeficiency virus [HIV], positive hepatitis B surface antigen (HBsAg), or positive hepatitis C virus [HCV] antibody
7. Subjects who are employees or immediate relatives of the employees of the Sponsor, any of its affiliates or partners, or of the clinical research study site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2016-12; Primary Completion 2017-11 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Site 744, Birmingham, Alabama
  - Site 727, Phoenix, Arizona
  - Site 723, Little Rock, Arkansas
  - Site 718, Rogers, Arkansas
  - Site 709, Los Angeles, California
  - Site 708, Orange, California
  - Site 729, San Diego, California
  - Site 725, Santa Monica, California
  - Site 738, Simi Valley, California
  - Site 733, Upland, California
  - Site 726, Colorado Springs, Colorado
  - Site 735, DeLand, Florida
  - Site 711, Hialeah, Florida
  - Site 721, Jacksonville, Florida
  - Site 740, Blue Ridge, Georgia
  - Site 720, Decatur, Georgia
  - Site 734, West Des Moines, Iowa
  - Site 739, Prairie Village, Kansas
  - Site 713, Wichita, Kansas
  - Site 706, Shreveport, Louisiana
  - Site 712, Baltimore, Maryland
  - Site 703, Boston, Massachusetts
  - Site 730, New Bedford, Massachusetts
  - Site 704, Minneapolis, Minnesota
  - Site 736, Hazelwood, Missouri
  - Site 737, Springfield, Missouri
  - Site 745, Las Vegas, Nevada
  - Site 716, Berlin, New Jersey
  - Site 746, Amherst, New York
  - Site 705, Manhattan, New York
  - Site 743, Williamsville, New York
  - Site 715, Raleigh, North Carolina
  - Site 728, Cincinnati, Ohio
  - Site 707, Dayton, Ohio
  - Site 701, Oklahoma City, Oklahoma
  - Site 741, Salem, Oregon
  - Site 717, Media, Pennsylvania
  - Site 731, Philadelphia, Pennsylvania
  - Site 742, Lincoln, Rhode Island
  - Site 710, Anderson, South Carolina
  - Site 724, Chattanooga, Tennessee
  - Site 719, Austin, Texas
  - Site 702, Plano, Texas
  - Site 714, Virginia Beach, Virginia
  - Site 722, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication of study results — https://pubmed.ncbi.nlm.nih.gov/31647577/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects who received placebo
- DFN-15: Subjects who received DFN-15
Period: Double-blind Period 1 (DB1)
Arm/Group | Placebo | DFN-15
Started (Randomized in DB1) | 311 | 311
Not Completed | 43 (2 subjects were randomized who were neither recorded as having completed nor discontinued DB1) | 42 (4 subjects were randomized who were neither recorded as having completed nor discontinued DB1)
Completed (Completed DB1) | 266 | 265
Not Completed | 45 | 46
Period: Double-blind Period 2 (DB2)
Arm/Group | Placebo | DFN-15
Started (Randomized in DB2) | 278 | 267
Not Completed | 16 (There is a 13 subject discrepancy that is accounted for by erroneous randomization entries and subjects who were randomized but not dosed in DB2.) | 20 (There is a 5 subject discrepancy that is accounted for by erroneous randomization entries and subjects who were randomized but not dosed in DB2.)
Completed (Completed DB2) | 249 | 242
Not Completed | 29 | 25

BASELINE CHARACTERISTICS:
Population: Baseline characteristics list the safety population (i.e., all subjects who were dosed during DB1). Note that there are 2 subjects in the placebo group and 2 subjects in the DFN-15 group, for whom no postdose efficacy data were collected. These individuals are, therefore, included in the baseline subject counts but are not included subsequent results reporting.
Groups:
- DB1 Placebo: Subjects received placebo in the Double-blind period 1 (DB1)
- DB1 DFN-15: Subjects received DFN-15 in the Double-blind period 1 (DB1)
- Total: Total of all reporting groups
Arm/Group | DB1 Placebo | DB1 DFN-15 | Total
Number analyzed (Participants) | 282 | 285 | 567
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.59) | 40.5 (11.68) | 40.3 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 252 | 494
  Male | 40 | 33 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 40 | 78
  Not Hispanic or Latino | 243 | 242 | 485
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 50 | 75 | 125
  White | 219 | 198 | 417
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are Pain-free at 2 Hours Postdose (DB1)
Description: Percentage of subjects who were pain-free 2 hours postdose compared between DFN-15 and placebo in the DB1 period (defined as a reduction from predose moderate [Grade 2] or severe [Grade 3] pain to none [Grade 0]) during DB1.
Time Frame: 2 hours post dose
Population: Full Analysis Set 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Placebo LOCF: Placebo - last observation carried forward (LOCF)
- DFN-15 LOCF: DFN-15 - last observation carried forward (LOCF)
- Placebo OC: Placebo - observed cases (OC)
- DFN-15 OC: DFN-15 - observed cases (OC)
Arm/Group | Placebo LOCF | DFN-15 LOCF | Placebo OC | DFN-15 OC
Number analyzed (Participants) | 280 | 283 | 280 | 283
percentage of subjects | 21.7 [16.8 to 27.1] | 35.6 [30.0 to 41.6] | 22.1 [17.2 to 27.7] | 35.8 [30.1 to 41.8]
Statistical Analysis 1: Comparison: Placebo LOCF vs DFN-15 LOCF; Last Observation Carried Forward (LOCF); Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.36 to 2.94]
Statistical Analysis 2: Comparison: Placebo OC vs DFN-15 OC; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.34 to 2.89]

2. Primary Outcome: Percentage of Subjects Who Are Free From Their MBS at 2 Hours Postdose (DB1)
Description: Percentage of subjects who are free from their most bothersome symptom (MBS) among nausea, photophobia, and phonophobia at 2 hours postdose during DB1.
Time Frame: 2 hours post dose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo LOCF | DFN-15 LOCF | Placebo OC | DFN-15 OC
Number analyzed (Participants) | 232 | 232 | 227 | 228
percentage of subjects | 44.8 [38.3 to 51.5] | 57.8 [51.1 to 64.2] | 45.4 [38.8 to 52.1] | 58.3 [51.6 to 64.8]
Statistical Analysis 1: Comparison: Placebo LOCF vs DFN-15 LOCF; last observation carried forward (LOCF); Test type: Superiority; p = 0.007, Fisher Exact; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.17 to 2.43]
Statistical Analysis 2: Comparison: Placebo OC vs DFN-15 OC; observed cases (OC); Test type: Superiority; p = 0.007, Fisher Exact; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.16 to 2.44]

3. Secondary Outcome: Freedom From Nausea, Photophobia, and Phonophobia Postdose (DB1 and DB2)
Description: The percentage of subjects who were free from nausea, photophobia, and phonophobia at 15, 30, and 45 minutes and 1, 1.5, 2, 4, and 24 hours postdose during each DB treatment period were summarized by symptom, treatment group, and time point.
Time Frame: 15 minutes through 24 hours
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- DB1 Placebo (Nausea): Placebo in 1st double-blind treatment phase (DB1) who were nausea free
- DB1 DFN-15 (Nausea): DFN-15 in 1st double-blind treatment phase (DB1) who were nausea free
- DB1 Placebo (Photophobia): Placebo in 1st double-blind treatment phase (DB1) who were photophobia free
- DB1 DFN-15 (Photophobia): DFN-15 in 1st double-blind treatment phase (DB1) who were photophobia free
- DB1 Placebo (Phonophobia): Placebo in 1st double-blind treatment phase (DB1) who were phonophobia free
- DB1 DFN-15 (Phonophobia): DFN-15 in 1st double-blind treatment phase (DB1) who were phonophobia free
- DB2 Placebo (Nausea): Placebo in 2nd double-blind treatment phase (DB2) who were nausea free
- DB2 DFN-15 (Nausea): DFN-15 in 2nd double-blind treatment phase (DB2) who were nausea free
- DB2 Placebo (Photophobia): Placebo in 2nd double-blind treatment phase (DB2) who were photophobia free
- DB2 DFN-15 (Photophobia): DFN-15 in 2nd double-blind treatment phase (DB2) who were photophobia free
- DB2 Placebo (Phonophobia); DB2 DFN-15 (Phonophobia): DFN-15 in 2nd double-blind treatment phase (DB2) who were phonophobia free
Arm/Group | DB1 Placebo (Nausea) | DB1 DFN-15 (Nausea) | DB1 Placebo (Photophobia) | DB1 DFN-15 (Photophobia) | DB1 Placebo (Phonophobia) | DB1 DFN-15 (Phonophobia) | DB2 Placebo (Nausea) | DB2 DFN-15 (Nausea) | DB2 Placebo (Photophobia) | DB2 DFN-15 (Photophobia) | DB2 Placebo (Phonophobia) | DB2 DFN-15 (Phonophobia)
Number analyzed (Participants) | 151 | 149 | 243 | 238 | 203 | 195 | 124 | 108 | 208 | 202 | 157 | 169
percentage of subjects
  15 minutes postdose | 16.8 [10.8 to 24.3] | 15.7 [10.0 to 23.0] | 8.8 [5.4 to 13.5] | 9.6 [5.9 to 14.4] | 15.7 [10.7 to 21.9] | 10.5 [6.4 to 16.1] | 14.5 [8.5 to 22.5] | 13.7 [7.7 to 22.0] | 7.5 [4.2 to 12.2] | 8.0 [4.6 to 12.9] | 8.5 [4.5 to 14.4] | 10.3 [6.0 to 16.1]
  30 minutes postdose | 33.6 [25.9 to 41.9] | 32.9 [25.3 to 41.1] | 13.0 [9.0 to 18.1] | 20.1 [15.1 to 25.9] | 26.0 [20.0 to 32.9] | 24.6 [18.6 to 31.4] | 26.9 [19.2 to 35.8] | 31.4 [22.7 to 41.2] | 14.4 [9.8 to 20.0] | 21.9 [16.4 to 28.4] | 15.6 [10.2 to 22.3] | 27.4 [20.8 to 34.9]
  45 minutes postdose | 43.8 [35.6 to 52.3] | 45.3 [37.1 to 53.7] | 20.2 [15.2 to 25.9] | 30.6 [24.7 to 37.0] | 26.7 [20.6 to 33.5] | 35.8 [29.0 to 43.0] | 41.8 [32.9 to 51.1] | 44.3 [34.7 to 54.3] | 22.1 [16.6 to 28.4] | 36.2 [29.5 to 43.3] | 25.8 [19.1 to 33.4] | 38.6 [31.1 to 46.4]
  1 hour postdose | 49.3 [41.0 to 57.7] | 56.8 [48.4 to 64.9] | 26.5 [21.0 to 32.6] | 38.9 [32.6 to 45.5] | 38.3 [31.4 to 45.5] | 45.0 [37.8 to 52.4] | 52.5 [43.2 to 61.6] | 51.9 [42.0 to 61.7] | 27.9 [21.9 to 34.6] | 43.7 [36.7 to 50.9] | 34.2 [26.8 to 42.2] | 44.0 [36.3 to 51.9]
  1.5 hours postdose | 58.5 [50.1 to 66.6] | 63.5 [55.2 to 71.3] | 36.0 [29.9 to 42.5] | 47.4 [40.9 to 54.0] | 47.2 [40.1 to 54.4] | 50.8 [43.5 to 58.1] | 60.2 [50.9 to 68.9] | 67.3 [57.5 to 76.0] | 35.4 [28.9 to 42.4] | 52.5 [45.3 to 59.6] | 43.2 [35.3 to 51.4] | 56.3 [48.4 to 63.9]
  2 hours postdose | 62.2 [53.8 to 70.0] | 67.6 [59.4 to 75.0] | 44.4 [37.9 to 50.9] | 58.3 [51.7 to 64.7] | 54.5 [47.3 to 61.5] | 61.1 [53.9 to 68.1] | 66.9 [57.9 to 75.1] | 69.2 [59.5 to 77.7] | 45.9 [39.0 to 52.9] | 64.0 [56.9 to 70.6] | 48.7 [40.6 to 56.8] | 67.7 [60.0 to 74.7]
  4 hours postdose | 75.5 [67.8 to 82.1] | 75.0 [67.2 to 81.7] | 61.2 [54.7 to 67.3] | 69.9 [63.6 to 75.7] | 72.9 [66.2 to 78.9] | 71.5 [64.6 to 77.8] | 74.2 [65.6 to 81.6] | 85.0 [76.9 to 91.2] | 62.8 [55.8 to 69.4] | 78.1 [71.7 to 83.6] | 59.0 [50.8 to 66.8] | 76.2 [69.0 to 82.4]
  24 hours postdose | 91.4 [85.7 to 95.3] | 90.6 [84.7 to 94.8] | 85.2 [80.1 to 89.4] | 85.7 [80.6 to 89.9] | 89.7 [84.6 to 93.5] | 85.1 [79.3 to 89.8] | 87.1 [79.9 to 92.4] | 93.5 [87.1 to 97.4] | 84.6 [79.0 to 89.2] | 91.6 [86.9 to 95.0] | 81.5 [74.6 to 87.3] | 90.5 [85.1 to 94.5]

4. Secondary Outcome: Time to Headache Pain Relief Postdose (DB1 and DB2)
Time Frame: 2 hours postdose
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Placebo DB1: Subjects received placebo in the 1st randomized double blind phase (DB1)
- DFN-15 DB1: Subjects received DFN-15 in the 1st randomized double blind phase (DB1)
- Placebo DB2: Subjects received placebo in the 2nd randomized double blind phase (DB2)
- DFN-15 DB2: Subjects received DFN-15 in the 2nd randomized double blind phase (DB2)
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
minutes | 59.5 (29.82) | 68.9 (43.67) | 55.3 (29.22) | 62.1 (29.58)

5. Secondary Outcome: Time to Headache Pain Freedom Postdose (DB1 and DB2)
Time Frame: 2 hours postdose
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 17 | 27 | 22 | 26
minutes | 66.6 (32.31) | 68.5 (31.01) | 68.8 (25.06) | 80.8 (25.80)

6. Secondary Outcome: Headache Pain Relief Postdose (DB1 and DB2)
Description: Headache pain relief during postdose in DB1 was defined as a reduction from moderate or severe pain at predose reduced to mild or none postdose, and for DB2 as moderate or severe pain at predose reduced to mild or none postdose, or mild pain at predose reduced to none postdose. Outcome measure shows percentage of subjects experiencing headache pain relief by time point.
Time Frame: 15 minutes to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects
  15 minutes postdose | 16.6 [12.1 to 22.0] | 13.4 [9.4 to 18.3] | 10.9 [7.1 to 15.8] | 11.7 [7.8 to 16.6]
  30 minutes postdose | 28.9 [23.4 to 34.9] | 32.2 [26.6 to 38.2] | 27.5 [21.9 to 33.7] | 31.6 [25.7 to 38.0]
  45 minutes postdose | 40.2 [34.2 to 46.5] | 46.5 [40.4 to 52.6] | 37.1 [31.0 to 43.5] | 47.7 [41.2 to 54.2]
  1 hour postdose | 45.1 [38.9 to 51.4] | 56.8 [50.7 to 62.7] | 43.8 [37.4 to 50.3] | 56.1 [49.5 to 62.5]
  1.5 hours postdose | 55.2 [48.9 to 61.4] | 70.0 [64.1 to 75.3] | 53.3 [46.8 to 59.7] | 66.4 [60.0 to 72.4]
  2 hours postdose | 60.5 [54.3 to 66.4] | 74.5 [69.0 to 79.6] | 60.7 [54.2 to 66.8] | 74.4 [68.3 to 79.8]
  4 hours postdose | 75.2 [69.5 to 80.3] | 79.6 [74.4 to 84.2] | 75.0 [69.1 to 80.3] | 82.2 [77.5 to 87.4]
  24 hours postdose | 92.5 [88.7 to 95.4] | 92.4 [88.7 to 95.3] | 89.0 [84.4 to 92.6] | 93.8 [89.9 to 96.5]

7. Secondary Outcome: Headache Pain Freedom Postdose (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 15, 30, and 45 minutes and 1, 1.5, 2 (DB2), and 4, and 24 hours postdose during each DB treatment period were summarized by treatment group.
Time Frame: 15 minutes to 24 hours postdose
Population: Data were not collected at 2 hours postdose during DB1 per protocol
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects
  15 minutes postdose | 1.3 [0.3 to 3.7] | 0.4 [0.0 to 2.2] | 1.4 [0.3 to 3.9] | 0.9 [0.1 to 3.2]
  30 minutes postdose | 3.6 [1.6 to 6.6] | 3.0 [1.3 to 5.8] | 6.4 [3.6 to 10.3] | 6.8 [4.0 to 10.9]
  45 minutes postdose | 8.6 [5.5 to 12.7] | 11.1 [7.6 to 15.4] | 11.7 [7.9 to 16.4] | 12.7 [8.7 to 17.6]
  1 hour postdose | 12.8 [9.0 to 17.6] | 17.9 [13.6 to 23.0] | 15.8 [11.5 to 21.1] | 23.2 [18.0 to 29.1]
  1.5 hours postdose | 17.4 [13.0 to 22.5] | 27.1 [21.9 to 32.8] | 25.2 [19.9 to 31.2] | 36.1 [30.0 to 42.6]
  2 hours postdose: number analyzed (Participants) | 0 | 0 | 248 | 243
  2 hours postdose |  |  | 31.1 [25.4 to 37.4] | 46.2 [39.8 to 52.8]
  4 hours postdose | 44.4 [38.3 to 50.6] | 56.4 [50.3 to 62.3] | 50.0 [43.6 to 56.4] | 61.9 [55.4 to 68.1]
  24 hours postdose | 77.2 [71.7 to 82.1] | 77.3 [72.0 to 82.1] | 75.1 [69.2 to 80.4] | 82.9 [77.5 to 87.5]

8. Secondary Outcome: Absence of Screening MBS at Time Points Postdose (DB1 and DB2)
Description: The percentage of subjects with their Screening MBS (most bothersome symptoms) among nausea, photophobia, and phonophobia (from eDiary data collection) absent at 15, 30, and 45 minutes and 1, 1.5, 2 (DB2 period), 4, and 24 hours postdose during each DB treatment period were summarized by treatment group and time point.
Time Frame: 15 minutes to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects
  15 minutes postdose | 10.6 [6.8 to 15.6] | 6.3 [3.4 to 10.5] | 8.0 [4.4 to 13.1] | 8.9 [5.2 to 14.1]
  30 minutes postdose | 17.4 [12.7 to 23.0] | 17.3 [12.6 to 22.9] | 15.8 [10.9 to 21.8] | 22.9 [17.1 to 29.5]
  45 minutes postdose | 22.5 [17.2 to 28.5] | 28.5 [22.7 to 34.8] | 27.5 [21.3 to 34.3] | 36.8 [30.0 to 44.1]
  1 hour postdose | 25.0 [19.5 to 31.1] | 39.6 [33.2 to 46.2] | 35.8 [29.0 to 43.0] | 44.7 [37.5 to 52.1]
  1.5 hours postdose | 38.7 [32.4 to 45.3] | 49.1 [42.5 to 55.8] | 42.6 [35.5 to 49.8] | 53.4 [46.1 to 60.6]
  2 hours postdose | 44.8 [38.3 to 51.5] | 57.8 [51.1 to 64.2] | 50.0 [42.8 to 57.2] | 63.4 [56.1 to 70.2]
  4 hours postdose | 61.3 [54.7 to 67.5] | 67.4 [61.0 to 73.4] | 60.7 [53.5 to 67.6] | 78.0 [71.5 to 83.7]
  24 hours postdose | 86.0 [80.9 to 90.2] | 82.5 [77.0 to 87.1] | 83.7 [77.7 to 88.6] | 89.6 [84.4 to 93.5]

9. Secondary Outcome: Change in Functional Disability Score Postdose (DB1 and DB2)
Description: The values of the functional disability scale were: 0=no disability, able to function normally; 1=performance of daily activities mildly impaired, can still do everything but with difficulty; 2=performance of daily activities moderately impaired, unable to do some things; 3=performance of daily activities severely impaired, cannot do all or most things, bed rest may be necessary.
  A decrease in values indicates improvement from baseline.
Time Frame: 2 to 24 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
units on a scale
  2 hours postdose | -0.7 (0.94) | -0.9 (1.00) | -0.6 (0.83) | -0.9 (0.87)
  4 hours postdose | -1.1 (0.99) | -1.3 (1.01) | -1.0 (0.95) | -1.2 (0.94)
  24 hours postdose | -1.8 (0.82) | -1.7 (0.84) | -1.5 (0.86) | -1.5 (0.88)

10. Secondary Outcome: Headache Pain Freedom Among Subjects With Cutaneous Allodynia (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 2 and 4 hours postdose during each DB treatment period among those subjects reporting cutaneous allodynia before dosing were summarized by treatment group and time point.
Time Frame: 2 to 4 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects
  2 hours postdose | 19.2 [9.6 to 32.5] | 38.0 [24.7 to 52.8] | 31.0 [17.6 to 47.1] | 54.3 [39.0 to 69.1]
  4 hours postdose | 45.3 [31.6 to 59.6] | 56.0 [41.3 to 70.0] | 40.5 [25.6 to 56.7] | 56.5 [41.1 to 71.1]

11. Secondary Outcome: Headache Pain Freedom Among BMI Category (DB1 and DB2)
Description: The percentage of subjects who were pain-free at 2 and 4 hours postdose whose BMI was <30 kg/m2 vs. subjects whose BMI was ≥30 kg/m2 during each DB treatment period were summarized by treatment group and time point.
Time Frame: 2 to 4 hours postdose
Population: Subjects were striated by BMI by dosing assignment for DB1 and DB2, therefore subject numbers differ from overall totals.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects
  2 hours postdose (BMI<30): number analyzed (Participants) | 150 | 146 | 142 | 117
  2 hours postdose (BMI<30) | 22.1 [15.8 to 29.7] | 31.5 [24.1 to 39.7] | 26.8 [19.7 to 34.8] | 41.9 [32.8 to 51.4]
  4 hours postdose (BMI <30): number analyzed (Participants) | 152 | 146 | 142 | 118
  4 hours postdose (BMI <30) | 41.7 [33.8 to 50.0] | 55.9 [47.4 to 64.1] | 50.0 [41.5 to 58.5] | 67.8 [58.6 to 76.1]
  2 hours postdose (BMI>=30): number analyzed (Participants) | 114 | 129 | 102 | 121
  2 hours postdose (BMI>=30) | 21.1 [14.0 to 29.7] | 40.3 [31.8 to 49.3] | 37.3 [27.9 to 47.4] | 50.4 [41.2 to 59.6]
  4 hours postdose (BMI>=30): number analyzed (Participants) | 115 | 130 | 102 | 121
  4 hours postdose (BMI>=30) | 47.8 [38.4 to 57.3] | 56.9 [48.0 to 65.6] | 50.0 [39.9 to 60.1] | 56.2 [46.9 to 65.2]

12. Secondary Outcome: Headache Pain Recurrence Postdose (DB1 and DB2)
Description: Headache pain recurrence was defined as pain-free at 2 hours postdose with pain reported as mild, moderate, or severe at 24 hours postdose. This outcome measure shows percentage of subjects who reported pain-free status and 2 hours postdose but subsequently reported recurrent pain at 24 hours postdose.
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects | 14.0 [6.3 to 25.8] | 9.2 [4.3 to 16.7] | 6.6 [2.2 to 14.7] | 6.4 [2.6 to 12.7]

13. Secondary Outcome: Sustained Headache Pain Relief Postdose (DB1 and DB2)
Description: Sustained headache pain relief was defined as pain relief at 2 hours postdose with no use of rescue medication and no worsening of headache pain within 2 to 24 hours postdose. This outcome measure shows the percentage of subjects who reported pain relief at 2 hours postdose with no use of rescue medication or worsening of headache pain through 24 hours postdose.
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects | 43.4 [36.6 to 50.4] | 55.1 [48.0 to 62.1] | 49.7 [42.4 to 57.1] | 60.2 [52.8 to 67.3]

14. Secondary Outcome: Sustained Headache Pain Freedom Postdose (DB1 and DB2)
Description: Sustained headache pain freedom was defined as pain-free at 2 hours postdose, with no use of rescue medication and no recurrence of headache pain within 2 to 24 hours postdose. This outcome measure shows percentage of subjects who were pain-free at 2 hours postdose without the use of rescue medication or recurrence of headache pain through 24 hours postdose.
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects | 17.0 [12.2 to 22.7] | 26.8 [20.9 to 33.4] | 26.5 [20.3 to 33.3] | 39.8 [32.7 to 47.2]

15. Secondary Outcome: Use of Rescue Medication Postdose (DB1 and DB2)
Description: The percentage of subjects who used rescue mediation after 2 hours (2 to 24 hours) postdose compared between DFN-15 and placebo in each DB period.
Time Frame: 2 to 24 hours postdose
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
percentage of subjects | 30.1 [24.7 to 36.0] | 15.8 [11.7 to 20.7] | 18.4 [13.7 to 23.8] | 16.7 [12.2 to 22.0]

16. Secondary Outcome: Subject-Rated Treatment Satisfaction Postdose (DB1 and DB2)
Description: Subject-rated treatment overall satisfaction was based on a 7-point scale at 2 and 4 hours postdose during each DB treatment period. The difference between the subject-rated study drug treatment satisfaction score at 2 and 4 hours postdose and the baseline PPMQ-R (Patient Perception of Migraine Questionnaire) response for the same question were summarized by treatment group (global satisfaction item at baseline asked about the subject's usual migraine treatment). The possible values of the subject treatment satisfaction scale were: 1=very satisfied, 2=satisfied, 3=somewhat satisfied, 4=neither satisfied nor dissatisfied, 5=somewhat dissatisfied, 6=dissatisfied, 7=very dissatisfied.
  A decrease in values indicates improvement from baseline.
Time Frame: 2 to 4 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 287 | 248 | 243
units on a scale
  2 hours postdose | 3.9 (1.90) | 3.3 (1.78) | 3.6 (1.97) | 3.1 (1.85)
  4 hours postdose | 3.7 (2.05) | 3.2 (1.90) | 3.5 (2.06) | 2.9 (1.80)

17. Secondary Outcome: Subject-Rated Treatment Satisfaction at 24 Hours Postdose - PPMQ-R (DB1 and DB2)
Description: Patient Perception of Migraine Questionnaire-Revised had 30 questions assessing subject's satisfaction with migraine medication, including 3 global items & 4 subscales (i.e., efficacy, function, ease of use, tolerability). A 5-point scale (1-Not At All to 5-Extremely) was used for tolerability subscale questions; a 7-point scale (1-Very Satisfied to 7-Very Dissatisfied) was used for all other subscales and global items. Total score was average of efficacy/function/ease of use subscale scores. Each subscale & total scores were transformed to range from 0-100, with higher scores indicating better satisfaction or tolerability. Total raw score/global items were not transformed. The total raw score could range from 17 (min) to 119 (max), with lower scores indicating better satisfaction. Change from baseline scores at 24-hour-postdose for each subscale score, global item score, total score, & total raw score were summarized by treatment group below.
Time Frame: 24 hours postdose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2
Number analyzed (Participants) | 280 | 283 | 248 | 243
units on a scale
  Total Score | -0.657 (30.9929) | 4.367 (33.7146) | 3.544 (32.3791) | 3.940 (31.7753)
  Total Raw Score | 0.835 (12.0599) | -1.254 (12.9334) | -0.744 (12.3973) | -1.448 (12.3105)
  Efficacy | -4.196 (39.0051) | 2.292 (40.8958) | 0.385 (39.7293) | 3.604 (39.9214)
  Function | -0.020 (40.3093) | 7.931 (42.8913) | 6.239 (39.8213) | 8.169 (38.6639)
  Ease of Use | 2.247 (28.5348) | 2.876 (29.3816) | 4.009 (28.6588) | 0.047 (28.8880)
  Tolerability | 5.99 (16.521) | 8.45 (15.930) | 9.01 (15.301) | 6.72 (15.565)
  Medication Effectiveness (Global Item) | 0.7 (2.59) | 0.2 (2.77) | 0.2 (2.64) | 0.2 (2.63)
  Side Effects (Global Item) | -0.3 (2.05) | 2.6 (1.36) | -0.7 (1.88) | -0.3 (1.92)
  Overall Satisfaction (Global Item) | 0.5 (2.67) | 0.1 (2.75) | 0.1 (2.62) | 0.0 (2.48)

ADVERSE EVENTS:
Time Frame: Per protocol, the maximum dosing timeframe for DB2 was 10 weeks; therefore, the maximum AE collection window was 11 weeks total.
Description: For DB1: TEAE that started or worsening of a pre-existing condition on or after the first dose of study drug (DFN-15 or placebo) in to taking DB2 study drug, whichever occurs first.
  For DB2: TEAE that started or worsened on or after the first dose of study drug in DB2 up to 5 days after the date of the last dose of study drug in DB2.
  Overall group includes all subjects who received at least one dose of study drug (DFN-15 or placebo) during DB1.
Groups:
- Placebo DB1: TEAEs that occurred following placebo dose in DB1
- DFN-15 DB1: TEAEs that occurred following DFN-15 dose in DB1
- Placebo DB2: TEAEs that occurred following placebo dose in DB2
- DFN-15 DB2: TEAEs that occurred following DFN-15 dose in DB2
- Overall: TEAEs that occurred following the first dose of placebo or DFN-15
Arm/Group | Placebo DB1 | DFN-15 DB1 | Placebo DB2 | DFN-15 DB2 | Overall
All-Cause Mortality (participants affected / at risk) | 0/282 | 0/285 | 0/249 | 0/244 | 0/567
Serious Adverse Events (participants affected / at risk) | 2/282 | 0/285 | 0/249 | 0/244 | 2/567
Other Adverse Events (participants affected / at risk) | 9/282 | 17/285 | 5/249 | 6/244 | 37/567
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo DB1 (N=282) | DFN-15 DB1 (N=285) | Placebo DB2 (N=249) | DFN-15 DB2 (N=244) | Overall (N=567)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo DB1 (N=282) | DFN-15 DB1 (N=285) | Placebo DB2 (N=249) | DFN-15 DB2 (N=244) | Overall (N=567)
Nausea (Gastrointestinal disorders) | 5 | 9 | 3 | 2 | 19
Dysgeusia (Nervous system disorders) | 4 | 12 | 2 | 4 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT03006276/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03006276/SAP_001.pdf